CLINICAL TRIAL: NCT01066325
Title: Improving Flexibility With a Mindbody Approach
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Parker Research Institute (Other)
Responsible Party: Principal Investigator, Dr. Anne M. Jensen, Research Faculty, Parker Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Sit-n-Reach Study
Record Dates: First submitted 2010-02-09; First posted 2010-02-10 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: General Low Back Hip and Hamstring Flexibility
Keywords: Sit-n-Reach Test; Flexibility; Hamstring; Mindbody; Complementary and Alternative Medicine; Neuro Emotional Technique (NET)

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- NET (Experimental): This arm will receive two 20-minutes sessions of NET 1 week apart. NET (Neuro Emotional Technique) is a non-invasive stress reduction technique.
  Interventions: Behavioral: Neuro Emotional Technique
- Active Controls (Active Comparator): This arm will receive two 20-minute sessions of stretching instructions 1 week apart.
  Interventions: Other: Stretching Instruction
- Inactive Controls (No Intervention): This arm will receive no intervention and no instructions.

INTERVENTIONS:
Behavioral: Neuro Emotional Technique — NET is considered an alternative stress-reduction technique. Its aim is to remove neurological abnormalities which have a specified physiopathological pattern. The goal of NET is to normalize the aberrant patterns through a physical correction.
  During the NET procedure, various psychological components of the anxious state are considered: cognitions, emotions, and behaviours. These various components are explored for a physiological reaction in the participant. Once a physiological reaction is found, the practitioner helps the participant identify the specific emotion. The procedure is concluded when the patient no longer feels distress or discomfort. Following the intervention, patients frequently report feeling subjective relief.
  Arms: NET
Other: Stretching Instruction — This arm is the Active Control Arm and will receive two 20-minute sessions of Stretching Instructions. During these instructions, participants will hold stretches for not longer than 5 seconds, which in not likely to have any therapeutic effect.
  Arms: Active Controls

SUMMARY:
The objectives of this study are to investigate if Neuro Emotional Technique (NET) will impact back and leg flexibility over both the short-term and the long-term.

It is hypothesized that NET will improve flexibility and that these changes are durable.

DETAILED DESCRIPTION:
General flexibility is a key component of health, wellbeing and general physical conditioning. In fact, lack of flexibility has been associated with an increased risk of developing musculoskeletal injuries and underperformance.

It has been previously shown that a regular stretching routine will improve flexibility relatively quickly. However, when the routine is discontinued or when stretching is not performed regularly, flexibility is also quickly lost. Therefore, an alternative intervention with longer retention would be desirable.

The reason for reduced flexibility, or a shortened muscle length, can be multifactorial. Reduced flexibility can be due to physical causes, such as an acute injury or strength training. Likewise, mental factors, such as anxiety and stress, can also significantly contribute to muscle tension, thereby reducing flexibility. It has been previously shown that somatic symptoms of anxiety can be lessened by treating the psychological symptoms of anxiety. It has also been previously shown that Neuro Emotional Technique® (NET), a chiropractic stress-reduction technique, is effective at reducing stress. Therefore, I hypothesize that NET may be effective at improving general flexibility. Therefore, the aim of this study is to investigate if NET can improve flexibility in the short-term, and if so, if these changes are durable in the long term.

Participants of this study will be randomly divided into three arms: (1) Experimental Arm - which will receive two 20-minute sessions of NET, (2) Active Controls - which will receive two 20-minute sessions of stretching instructions, and (3) Inactive Control - which will receive no intervention or instruction, but simply be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 45 years.

Exclusion Criteria:

* A currently diagnosed physical or mental health problem
* Pain on forward bending
* Pregnancy

NOTE: For this study, no compensation is possible.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2010-03; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Change in Sit-n-Reach Test Scores (cm) | weeks 0, 3

SECONDARY OUTCOMES:
Depression, Anxiety and Stress Scales (DASS) score - change | weeks 0, 3

CONTACTS AND LOCATIONS:
Overall Officials: Anne M Jensen, DC, MS, MSc, Principal Investigator — Parker Research Institute
Locations (1):
- Parker Research Institute, Dallas, Texas, United States

REFERENCES:
- [Background] Witvrouw E, Danneels L, Asselman P, D'Have T, Cambier D. Muscle flexibility as a risk factor for developing muscle injuries in male professional soccer players. A prospective study. Am J Sports Med. 2003 Jan-Feb;31(1):41-6. doi: 10.1177/03635465030310011801. PMID 12531755
- [Background] Wells GD, Elmi M, Thomas S. Physiological correlates of golf performance. J Strength Cond Res. 2009 May;23(3):741-50. doi: 10.1519/JSC.0b013e3181a07970. PMID 19387406
- [Background] Jensen AM, Ramasamy A. Treating spider phobia using Neuro Emotional Technique: findings from a pilot study. J Altern Complement Med. 2009 Dec;15(12):1363-74. doi: 10.1089/acm.2008.0595. PMID 20001838
- [Background] Baltaci G, Un N, Tunay V, Besler A, Gerceker S. Comparison of three different sit and reach tests for measurement of hamstring flexibility in female university students. Br J Sports Med. 2003 Feb;37(1):59-61. doi: 10.1136/bjsm.37.1.59. PMID 12547745
- [Background] Castro-Pinero J, Chillon P, Ortega FB, Montesinos JL, Sjostrom M, Ruiz JR. Criterion-related validity of sit-and-reach and modified sit-and-reach test for estimating hamstring flexibility in children and adolescents aged 6-17 years. Int J Sports Med. 2009 Sep;30(9):658-62. doi: 10.1055/s-0029-1224175. Epub 2009 Jul 7. PMID 19585399
- [Background] Chung PK, Yuen CK. Criterion-related validity of sit-and-reach tests in university men in Hong Kong. Percept Mot Skills. 1999 Feb;88(1):304-16. doi: 10.2466/pms.1999.88.1.304. PMID 10214658
- [Background] Ortega FB, Artero EG, Ruiz JR, Vicente-Rodriguez G, Bergman P, Hagstromer M, Ottevaere C, Nagy E, Konsta O, Rey-Lopez JP, Polito A, Dietrich S, Plada M, Beghin L, Manios Y, Sjostrom M, Castillo MJ; HELENA Study Group. Reliability of health-related physical fitness tests in European adolescents. The HELENA Study. Int J Obes (Lond). 2008 Nov;32 Suppl 5:S49-57. doi: 10.1038/ijo.2008.183. PMID 19011654
- [Background] Youdas JW, Krause DA, Hollman JH. Validity of hamstring muscle length assessment during the sit-and-reach test using an inclinometer to measure hip joint angle. J Strength Cond Res. 2008 Jan;22(1):303-9. doi: 10.1519/JSC.0b013e31815f5b7d. PMID 18296990
- [Background] Crawford JR, Henry JD. The Depression Anxiety Stress Scales (DASS): normative data and latent structure in a large non-clinical sample. Br J Clin Psychol. 2003 Jun;42(Pt 2):111-31. doi: 10.1348/014466503321903544. PMID 12828802
- [Background] Khan RS, Marlow C, Head A. Physiological and psychological responses to a 12-week BodyBalance training programme. J Sci Med Sport. 2008 Jun;11(3):299-307. doi: 10.1016/j.jsams.2007.04.005. Epub 2007 Aug 14. PMID 17698412
- [Background] Monti DA, Stoner ME, Zivin G, Schlesinger M. Short term correlates of the Neuro Emotional Technique for cancer-related traumatic stress symptoms: a pilot case series. J Cancer Surviv. 2007 Jun;1(2):161-6. doi: 10.1007/s11764-007-0018-x. PMID 18648957
- [Background] Monti DA, Sinnott J, Marchese M, Kunkel EJ, Greeson JM. Muscle test comparisons of congruent and incongruent self-referential statements. Percept Mot Skills. 1999 Jun;88(3 Pt 1):1019-28. doi: 10.2466/pms.1999.88.3.1019. PMID 10407911
- [Background] Peterson KB. A preliminary inquiry into manual muscle testing response in phobic and control subjects exposed to threatening stimuli. J Manipulative Physiol Ther. 1996 Jun;19(5):310-6. PMID 8792320